CLINICAL TRIAL: NCT05035030
Title: An Open Label Study to Evaluate the Long-term Safety and Efficacy of Odevixibat (A4250) in Patients With Alagille Syndrome (ASSERT-EXT)
Brief Title: Long-term Safety and Efficacy of Odevixibat in Patients With Alagille Syndrome
Acronym: ASSERT-EXT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Albireo, an Ipsen Company (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4250-015; 2023-509028-17-00 (EU CTIS Number); 2021-000996-36 (EudraCT Number)
Record Dates: First submitted 2021-08-13; First posted 2021-09-05 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Alagille Syndrome
MeSH Terms: conditions — Alagille Syndrome | interventions — odevixibat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Odevixibat (A4250) (Experimental): Capsules for oral administration once daily for 72 weeks.
  Interventions: Drug: Odevixibat

INTERVENTIONS:
Drug: Odevixibat — Odevixibat is a small molecule and selective inhibitor of IBAT.
  Other Names: A4250

SUMMARY:
The purpose of this study is to assess the long-term safety and effectiveness of odevixibat in participants with Alagille syndrome (ALGS).

The participants of this study will have ALGS a rare genetic disorder that can affect multiple organ systems of the body including the liver, heart, skeleton, eyes and kidneys. Common symptoms, which often develop during the first three months of life, include blockage of the flow of bile from the liver (cholestasis), yellowing of the skin and mucous membranes (jaundice), poor weight gain and growth and severe itching (pruritis).

The drug used for the study is odevixibat and was authorized for the treatment of cholestatic pruritus in infants with ALGS over 12 months of age by the United States Food and Drug Administration on 13 June 2023.

DETAILED DESCRIPTION:
This Phase 3, open-label, multi-center extension study will have two groups of participants: Cohort 1 (participants who participated in Study A4250-012 [NCT04674761; ASSERT] and meet the entry criteria for this study) and Cohort 2 (infants under 12 months of age) with ALGS.

The study will consist of 2 or 3 periods:

1. A 'Treatment period' of 72 weeks (cohort 1) or 12 weeks (cohort 2). Participants will visit the clinic every 4 to 12 weeks and will receive a dose of 120 μg/kg odevixibat daily.
2. An 'Optional extension period' where participants who wish to continue receiving odevixibat after the 'treatment period' will have the opportunity to remain on treatment with visits every 16 weeks until the drug is commercially available. The optional extension is available provided continued use is supported by the risk-benefit profile, the participant has not been previously withdrawn or discontinued from the study, and the study is not terminated by the Sponsor.
3. A 'Safety follow-up period' of 4 weeks (cohort 1) or 2 weeks (cohort 2). The Safety Follow-up Period will not occur for those who remain on treatment in the optional extension period.

Participants will need to complete an e-diary and questionnaires throughout the study (cohort 1 only). Participants will undergo blood samplings, urine collections (cohort 1 only), physical examinations, and clinical evaluations. They may continue some other medications, but the details need to be recorded.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1 :

1. Completion of the 24-week Treatment Period of Study A4250-012
2. Signed informed consent and assent as appropriate. Patients who turn 18 years of age (or legal age per country) during the study will be required to re-consent to remain on the study
3. Caregivers (and age-appropriate patients) must be willing and able to use an electronic diary (eDiary) device as required by the study
4. Sexually active males and females must agree to use a reliable contraceptive method with ≤1% failure rate (such as hormonal contraception, intra-uterine device, or complete abstinence) from signed informed consent through 90 days after last dose of study drug.

Cohort 2 :

1. Infant with clinically confirmed ALGS , ≤11 months of age at Study Day 1
2. Body weight ≥2 kg at Study Day 1
3. Gestational age ≥36 weeks. For children born with gestational age between 32 and 36 weeks, a postmenstrual age of ≥36 weeks is required .
4. Signed parent/legal guardian informed consent.

Exclusion Criteria:

Cohort 1 :

1. Decompensated liver disease, history or presence of clinically significant ascites, variceal hemorrhage, and/or encephalopathy
2. Patients who were not compliant with study drug treatment or procedures in Study A4250-012
3. Any other conditions or abnormalities which, in the opinion of the investigator, may compromise the safety of the patient, or interfere with the patient participating in or completing the study
4. Known hypersensitivity to any components of odevixibat

Cohort 2 :

1. Patient with past medical history or ongoing presence of other types of liver disease including, but not limited to, the following:

   1. Biliary atresia of any kind
   2. Progressive familial intrahepatic cholestasis (PFIC)
   3. Benign recurrent intrahepatic cholestasis
2. Patient with a past medical history or ongoing presence of any other disease or condition known to interfere with the absorption, distribution, metabolism (specifically bile acid metabolism), or excretion of drugs in the intestine, including but not limited to, inflammatory bowel disease
3. Patient with past medical history or ongoing chronic diarrhea requiring intravenous fluid or nutritional intervention for treatment of the diarrhea and/or its sequelae
4. Patient has a confirmed past diagnosis of infection with human immunodeficiency virus or other present and active, clinically significant chronic infection
5. Recent infection requiring hospitalization or treatment with parenteral anti-infective within 4 weeks of Study Day 1 or completion of oral anti-infective treatment within 2 weeks prior to the Screening Visit
6. Cancer diagnosis (except for basal cell carcinoma)
7. Chronic kidney disease with an impaired renal function and a glomerular filtration rate <70 mL/min/1.73 m2
8. Patient with surgical history of disruption of the enterohepatic circulation (biliary diversion surgery) within 6 months prior to the Screening Visit
9. Patient has had a liver transplant, or a liver transplant is planned within 6 months of Study Day 1
10. Decompensated liver disease, history or presence of clinically significant ascites, variceal hemorrhage, and/or encephalopathy
11. International normalized ratio (INR) >1.4 (the patient may be treated with Vitamin K, and if INR is ≤1.4 at resampling the patient may be enrolled)
12. Serum alanine aminotransferase (ALT) >10 × upper limit of normal (ULN) at Screening
13. Serum ALT >15 × ULN at any time point during the last 6 months unless an alternate etiology was confirmed for the elevation
14. Total bilirubin >15 × ULN at Screening
15. Patient suffers from uncontrolled, recalcitrant pruritic condition other than ALGS. Examples include, but not limited to, refractory atopic dermatitis or other primary pruritic skin diseases.
16. Patient exposed to alcohol or substance abuse in utero
17. Bile acid or lipid binding resins and medications that slow gastrointestinal motility
18. Patient has had investigational exposure to a drug, biologic agent, or medical device within 30 days prior to the Screening Visit, or 5 half-lives of the study agent, whichever is longer
19. Any other conditions or abnormalities which, in the opinion of the investigator may compromise the safety of the patient, or interfere with the patient participating in or completing the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-09-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in pruritus | Baseline to week 72 (cohort 1).
  Assessed as change in scratching score as measured by measured by the Albireo Observer-Reported Outcome Caregiver Instrument.
Percentage of participants with Treatment Emergent Adverse Event (TEAEs) and Serious Adverse Events (SAEs) | Baseline to week 12 (cohort 2).
  An Adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A serious adverse event (SAE) is an AE that results in any of following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Treatment-emergent adverse events. TEAEs included both Serious TEAEs and non-serious TEAEs.
Percentage of participants with clinically significant changes from baseline in Physical Examination | Baseline to week 12 (cohort 2).
  The clinical significance will be graded by the investigator.
Percentage of participants with clinically significant changes in Laboratory Parameters | Baseline to week 12 (cohort 2).
  The following laboratory parameters will be reported: blood chemistry, hematology and coagulation. The clinical significance will be graded by the investigator.
Percentage of participants with clinically significant changes from baseline in Vital Signs. | Baseline to week 12 (cohort 2).
  The clinical significance will be graded by the investigator.
Change from baseline in concomitant medications. | Baseline to week 12 (cohort 2).
Change from baseline in fat-soluble vitamin levels. | Baseline to week 12 (cohort 2).

SECONDARY OUTCOMES:
Change from baseline in serum bile acids levels | Baseline to week 72 (cohort 1).
Change from baseline in patient reported and observer reported itching and scratching severity scores | Baseline to week 72 (cohort 1).
  Assessed by the the Albireo ObsRO/ Patient Reported Outcomes (PRO) instruments. The Albireo ObsRO/PRO scratching and itch severity items use 0 to 4 response scales, where each response is distinguished by a unique facial expression, verbal anchor, number, and color code.
Percentage of participants achieving a clinically meaningful decrease in pruritus (pruritus responders) | Baseline to week 72 (cohort 1).
  Assessed by the Albireo ObsRO/patient reported outcomes (PRO) instruments
Change from baseline in sleep parameters. | Baseline to week 72 (cohort 1).
  Assessed with the Albireo ObsRO/PRO instruments (e.g: tiredness and number of awakenings).
Change from baseline in Pediatric Quality of Life Inventory (PedsQL) scores. | Baseline to week 72 (cohort 1).
  The PedsQL instrument consists of 36 questions and uses a 5-point response scales, where higher scores indicates worst symptoms.
Change from baseline in in Global Symptom Relief: Patient Global Impression of Improvement (PGIC) score. | Baseline to Weeks 4, 12, 24, 48 and 72 (cohort 1).
  The Patient Global Impression of Change (PGIC) is a patient-reported instrument that measures change in overall status on a scale ranging from one ("very much improved") to seven ("very much worse").
Change from baseline in in Global Symptom Relief: Clinical Global Impression of Improvement (CGIC) score. | Baseline to Weeks 4, 12, 24, 48 and 72 (cohort 1).
  The Clinical Global Impression of Change (CGIC) is a clinician-reported instrument that measures change in overall status on a scale ranging from one ("very much improved") to seven ("very much worse").
Change from baseline in in Global Symptom Relief: Caregiver Global Impression of Change (CaGIC) score | Baseline to Weeks 4, 12, 24, 48 and 72 (cohort 1).
  The caregiver Global Impression of Change is a caregiver-reported instrument that measures change in overall status on a scale ranging from one ("very much improved") to seven ("very much worse").
Change from baseline in serum bile acid levels. | Baseline through week 72 (cohort 1).
Percentage of participants with Treatment Emergent Adverse Event (TEAEs) and Serious Adverse Events (SAEs) | Baseline to week 72 (cohort 1).
  An Adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A serious adverse event (SAE) is an AE that resultes in any of following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Treatment-emergent adverse events. TEAEs included both Serious TEAEs and non-serious TEAEs.
Number of participants with change from baseline in physical examination | Baseline to week 72 (cohort 1).
Number of participants with change from baseline in vital signs | Baseline to week 72 (cohort 1).
Change from baseline in concomitant medications | Baseline to week 72 (cohort 1).
Change from baseline in laboratory test results Pharmacokinetic (PK) Cmax [Time Frame: Day 1, Week 4, Week 8, and Week 12] | Baseline to week 72 (cohort 1).
Change from baseline in plasma concentration of study drug | Day 1, Week 4, Week 8, and Week 12 (cohort 1).
Pharmacodynamic Parameters: Change in serum bile acids levels | Baseline to Week 12 (cohort 2).

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (34):
- United States (17):
  - Rady Children's Hospital, San Diego, California
  - UCSF, San Francisco, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Riley Hospital for Children at IU Health, Indianapolis, Indiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Mercy Hospital and Clinics, Kansas City, Missouri
  - Northwell Health System, New Hyde Park, New York
  - Hassenfeld Children's Hospital at NYU Langone, New York, New York
  - The Childrens Hospital at Montefiore Albert Einstein School of Medicine, The Bronx, New York
  - Atrium Health Carolinas Medical, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Oregon Health Science University School of Medicine, Portland, Oregon
  - Monroe Carell Jr. Childrens Hospital at Vanderbilt, Nashville, Tennessee
  - Childrens Medical Center of Dallas University of Texas Southwestern, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Texas Liver Institute, San Antonio, Texas
- Cliniques Universitaires Saint-Luc Bruxelles, Brussels, Belgium
- France (3):
  - Hôpital Femme Mère Enfant de Lyon, Bron
  - Antenne pediatrique du CIC-Hopital Jeanne De Flandre, Lille
  - Hopital Necker Enfants Malades, Paris
- Germany (3):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Medizinische Hochschul, Hanover
  - Universitatsklinik fur Kinder-und Jugendmedizin Tubingen, Tübingen
- Italy (3):
  - AOU Meyer, Florence
  - Azienda Ospedale University, Padua
  - Ospedale Pediatrico Bambino Gesu, Rome
- University of Malaya Medical Center, Kuala Lumpur, Malaysia
- Netherlands (2):
  - Universitair Medisch Centrum Groningen, Groningen
  - Wilhelmina Children's Hospital UMCU Utrecht, Utrecht
- Instytut Pomnik-Centrum Zdrowia Dzieck, Warsaw, Poland
- Istanbul University Istanbul Medical Faculty Hospital, Istanbul, Turkey (Türkiye)
- United Kingdom (2):
  - Birmingham Women's and Children's NHS Foundation Trust, Birmingham
  - King's College Hospital NHS Foundation Trust King's College Hospital Paediatric Research, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/